CLINICAL TRIAL: NCT00073177
Title: A 24 Week, Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Oral Roflumilast (250 mcg or 500 mcg) Daily in Patients With Asthma
Brief Title: Efficacy and Safety of Roflumilast in Patients With Asthma (BY217/M2-012)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-012
Record Dates: First submitted 2003-11-17; First posted 2003-11-19 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The aim of the study is to compare the effects of oral roflumilast with placebo on lung function in patients with asthma.

ELIGIBILITY:
Main Inclusion Criteria:

* Persistent bronchial asthma
* No change in asthma treatment within 4 weeks prior to visit 1
* Non-smoker or ex-smoker (for 12 months or longer)

Main Exclusion Criteria:

* Poorly controlled asthma or seasonal asthma
* History of lower airway infection four weeks prior to visit 1
* Chronic obstructive pulmonary disease (COPD) and/or other relevant lung disease
* Patients using > 8-puffs/day-short-acting bronchodilator (beta-agonists) (more than 3 days per week on average) prior to visit 1
* Clinically relevant abnormal laboratory values suggesting an undiagnosed disease, severe renal insufficiency, active hepatitis or an HIV infection
* Diagnosis, treatment or remission of any cancer (other than basal cell carcinoma) within two years prior to visit 1
* Patients with chronic heart failure
* Suspected hypersensitivity and/or contraindication to roflumilast or albuterol/salbutamol
* Female patients of childbearing potential not using adequate means of birth control or pregnant or breast-feeding females
* Patients who have received any investigational medication or device in the month prior to visit 1 or who plan to use another investigational medication during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819
Dates: Start 2003-11

PRIMARY OUTCOMES:
change in lung function from baseline to final visit.

SECONDARY OUTCOMES:
pulmonary function variables
diary variables
quality of life variables
time to first exacerbation
number of asthma exacerbations
safety.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (41):
- United States (37):
  - ALTANA Pharma, Cities in Alabama, Alabama
  - ALTANA Pharma, Cities in Arizona, Arizona
  - ALTANA Pharma, Cities in Arkansas, Arkansas
  - ALTANA Pharma, Cities in California, California
  - ALTANA Pharma, Cities in Colorado, Colorado
  - ALTANA Pharma, Cities in Florida, Florida
  - ALTANA Pharma, Cities in Georgia, Georgia
  - ALTANA Pharma, Cities in Idaho, Idaho
  - ALTANA Pharma, Cities in Illinois, Illinois
  - ALTANA Pharma, Cities in Indiana, Indiana
  - ALTANA Pharma, Cities in Iowa, Iowa
  - ALTANA Pharma, Cities in Kansas, Kansas
  - ALTANA Pharma, Cities in Kentucky, Kentucky
  - ALTANA Pharma, Cities in Louisiana, Louisiana
  - ALTANA Pharma, Cities in Maryland, Maryland
  - ALTANA Pharma, Massachusetts, Massachusetts
  - ALTANA Pharma, Cities in Michigan, Michigan
  - ALTANA Pharma, Cities in Minnesota, Minnesota
  - ALTANA Pharma, Cities in Mississippi, Mississippi
  - ALTANA Pharma, Cities in Missouri, Missouri
  - ALTANA Pharma, Cities in Montana, Montana
  - ALTANA Pharma, Cities in Nebraska, Nebraska
  - ALTANA Pharma, Cities in Nevada, Nevada
  - ALTANA Pharma, Cities in New Jersey, New Jersey
  - ALTANA Pharma, Cities in New York, New York
  - ALTANA Pharma, Cities in North Carolina, North Carolina
  - ALTANA Pharma, Cities in North Dakota, North Dakota
  - ALTANA Pharma, Cities in Oregon, Oregon
  - ALTANA Pharma, Cities in Pennsylvania, Pennsylvania
  - ALTANA Pharma, Cities in Rhode Island, Rhode Island
  - ALTANA Pharma, Cities in South Carolina, South Carolina
  - ALTANA Pharma, Cities in Tennessee, Tennessee
  - ALTANA Pharma, Cities in Texas, Texas
  - ALTANA Pharma, Cities in Utah, Utah
  - ALTANA Pharma, Cities in Virginia, Virginia
  - ALTANA Pharma, Cities in Washington, Washington
  - ALTANA Pharma, Cities in Wisconsin, Wisconsin
- ALTANA Pharma, Cities in Argentina, Argentina
- ALTANA Pharma, Cities in Colombia, Colombia
- ALTANA Pharma, Cities in Mexico, Mexico
- ALTANA Pharma, Cities in Peru, Peru

REFERENCES:
- [Derived] Chervinsky P, Meltzer EO, Busse W, Ohta K, Bardin P, Bredenbroker D, Bateman ED. Roflumilast for asthma: Safety findings from a pooled analysis of ten clinical studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S28-34. doi: 10.1016/j.pupt.2015.11.003. Epub 2015 Nov 22. PMID 26612545
- [Derived] Meltzer EO, Chervinsky P, Busse W, Ohta K, Bardin P, Bredenbroker D, Bateman ED. Roflumilast for asthma: Efficacy findings in placebo-controlled studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S20-7. doi: 10.1016/j.pupt.2015.10.006. Epub 2015 Oct 21. PMID 26498386
- See also: BY217-M2-012-RDS-2007-01-02.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4471&filename=BY217-M2-012-RDS-2007-01-02.pdf